CLINICAL TRIAL: NCT01860144
Title: An Observational Study of Bevacizumab in Chinese Patients With Metastatic Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, Director of GI oncology, Peking University
Other Study IDs: CGOG2001
Record Dates: First submitted 2013-05-19; First posted 2013-05-22 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Metastatic Colorectal Cancer
Keywords: bevacizumab; overall survival; adverse events; tumor resection rate
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- bevacizumab: Patients with metastatic colorectal cancer who accept treatment with chemotherapy and bevacizumab
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab
  Other Names: avastin

SUMMARY:
This observational, multicenter, prospective study will evaluate the use of bevacizumab in real clinical practice in chinese patients with metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed metastatic colorectal cancer patients Having initiated treatment with bevacizumab

Exclusion Criteria:

* non-metastatic colorectal cancer patients not recieved bevacizumab

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: metastatic colorectal cancer patients accept bevacizumab
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2012-06; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 6 weeks
  To evaluate the treatment response of bevacizumab in Chinese patients with mCRC in real clinical practice

SECONDARY OUTCOMES:
overall survival | 3 months
  OS means that from the first dose of treatment drug to death or lost, the follow-up visit will be performed every 3 months till death or lost
progression free survival | 6 weeks
  the follow-up visit of PFS will be performed every 6 weeks
Proportion of patients with bevacizumab treatment discontinuation | 3 weeks
  Proportion of patients with bevacizumab treatment discontinuation due to bevacizumab-related adverse events
resection rate | 1 month
  resection rate of tumor after chemotherapy plus bevacizumab

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, M.D., Principal Investigator — Beijing Cancer Hopital
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China